CLINICAL TRIAL: NCT05301413
Title: Addressing Social Determinants of Health to Improve Diabetes Prevention Program Outcomes Among Underserved African Americans (FIT4ALL Project)
Brief Title: Social Determinants and a Diabetes Prevention Program Tailored for African Americans
Acronym: FIT4ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: University of Massachusetts, Amherst (Other); University of Kansas (Other); Children's Mercy Hospital Kansas City (Other); University Health (Unknown)
Responsible Party: Principal Investigator, Jannette Berkley-Patton, Professor, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2048442
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: PreDiabetes; Overweight and Obesity
Keywords: African American; Prediabetes; Diabetes Prevention Program; Cultural tailoring; Linkage to care; Weight loss; Class attendance
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (Active Comparator): Standard Diabetes Prevention Program (DPP)
  Interventions: Behavioral: Diabetes Prevention Program
- Culturally Tailored DPP (Experimental): DPP culturally tailored for African Americans
  Interventions: Behavioral: Culturally Tailored Diabetes Prevention Program; Behavioral: Diabetes Prevention Program
- Culturally Tailored DPP Enhanced with Socioeconomic Supports (Experimental): Culturally tailored DPP plus promotions for class attendance, hybrid attendance (in-person and virtual), and linkage to care services provided by a community health worker
  Interventions: Behavioral: Culturally Tailored Diabetes Prevention Program; Behavioral: Culturally Tailored DPP Enhanced with Socioeconomic Supports; Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Culturally Tailored Diabetes Prevention Program — This intervention includes a culturally tailored DPP curriculum, class procedures, and handouts
  Other Names: Culturally Tailored DPP
  Arms: Culturally Tailored DPP; Culturally Tailored DPP Enhanced with Socioeconomic Supports
Behavioral: Culturally Tailored DPP Enhanced with Socioeconomic Supports — This intervention includes the culturally tailored DPP curriculum, class procedures, and handouts along with promotional items for class participation, opportunities to attend class in-person or virtually through a digital platform, and assistance from a community health worker to provide linkage to health care services and community resources
  Other Names: FIT4ALL
  Arms: Culturally Tailored DPP Enhanced with Socioeconomic Supports
Behavioral: Diabetes Prevention Program — This is the CDC TD2 evidence-based Diabetes Prevention Program
  Other Names: DPP

SUMMARY:
African Americans (AAs) have rates of diabetes mellitus (DM) twice that of Whites and are disproportionately affected by leading risk factors for DM - obesity and low-income. A critical strategy in the battle against DM is the Diabetes Prevention Program (DPP), an evidence-based intervention that significantly delays or prevents Type 2 diabetes through the promotion of diet change, exercise and modest weight loss. However, weight loss from the DPP among AAs is about half that of White participants, and suboptimal AA attendance is a critical contributor. The investigators propose to conduct a study that will address social determinants (SD) that challenge DPP attendance with underserved African Americans from a safety net hospital. The investigators will examine DPP attendance and weight loss with participants randomized to 3 groups: standard DPP, a culturally-tailored DPP to address acceptability, and a culturally-tailored DPP enhanced to address socioeconomic-related barriers to DPP participation. This novel study is the first to tailor the DPP to address SD cultural and socioeconomic barriers that limit DPP attendance and reduce its effectiveness on outcomes. The proposed multidimensional, SD tailored DPP has great potential to be a feasible and scalable model to reduce DM risks among urban, African Americans and ultimately reduce DM disparities.

DETAILED DESCRIPTION:
African Americans (AAs) are disproportionately burdened by diabetes mellitus (DM) with rates twice as high as Whites (13% vs 7.5%), and increased rates of DM-related complications and comorbidities (e.g. amputations, cardiovascular disease). A key pre-DM risk factor is overweight/obesity. Nearly 70% of AAs are overweight or obese, with higher rates among AAs with low-income. A critical component of national efforts to reduce growing obesity rates and prevent DM is the Diabetes Prevention Program (DPP), a lifestyle intervention proven to reduce or delay DM onset with diet change, exercise, and modest weight loss (5-7%) in a rigorously evaluated national trial. A group-based version of the DPP has been widely disseminated and numerous community-based trials support its efficacy. In spite of these successes, there are significant health disparities in DPP attendance and outcomes and considerable room exists for improving success rates among AAs, a population that tends to experience half the amount of DPP weight loss compared to Whites. The investigators aim to build on our promising pilot studies by tailoring the DPP via a social determinants (SD) of health lens to achieve optimal DPP attendance and clinically meaningful weight loss with pre-DM AAs. This includes tailoring on cultural and socioeconomic SD mechanisms that are associated with improving health outcomes and align with predisposing needs among AAs who are primarily of low-income and live in low-resource AA communities.

The investigators propose a randomized controlled trial of 360 pre-DM AA patients from a safety net hospital (SNH) to test a standard DPP (S-DPP) against a culturally tailored DPP (TC-DPP; e.g., tailoring of language, foods, values, religiosity, norms, values) alone and a culturally tailored DPP enhanced to address access and support related economic barriers (TCE-DPP; hybrid group/online/text DPP; community health worker support to improve access to DPP classes, healthy food, exercise, and other community and health resources; and class promotions) over 12 months. The investigators will: 1) examine effects of TC-DPP and TCE-DDP on percent weight loss and attendance (primary outcomes) and on secondary outcomes (physical activity, completion of physician follow-up visit, hbA1c, and blood pressure) at 6 and 12 months with SNH AAs, 2) evaluate potential mediators/ moderators related to weight loss and attendance among AA SNH patients at 6 and 12 months to determine modifiable facilitators and barriers, and 3) conduct a process evaluation to examine TCE-DPP acceptability, feasibility, and fidelity, and relationships between delivery dose, exposure, costs, and outcomes to identify and improve essential intervention components. Our multidimensional DPP interventions are guided by our past pilots, and based on components that, all together, were used to help drive clinically important outcomes in the original DPP trial - and are certainly needed to achieve similar outcomes with AA primarily of low-income. To our knowledge this is the first study to test multidimensional tailoring via an SD lens to truly impact DPP attendance and outcomes, and has potential to be a feasible, scalable model to reduce DM disparities among at-risk AA.

ELIGIBILITY:
Inclusion Criteria:

* Black/African American
* Overweight ([BMI> 24); and
* Diagnosed with prediabetes OR pre-diagnosed with gestational diabetes OR high risk result on prediabetes risk test

Exclusion Criteria:

* Diagnosed with diabetes
* Pregnant
* Not fluent in English
* Currently pregnant, planning a pregnancy in the next year, currently breastfeeding or have given birth in the last 6 months
* Currently participating in a weight loss program
* Currently have a medical condition that causes drastic weight loss
* Bariatric weight loss surgery in last year
* Cannot walk a 1-block distance without assistance and without stopping due to pain, tightness, or pressure in the chest
* Had heart failure
* Not willing to use a fitness tracker, wi-fi scale, and the internet
* Not available in the evening one day each week to participate in a class

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Percent Weight Loss | 6 months
  Percentage of weight loss from initial baseline weight
Percent Weight Loss | 12 months
  Percentage of weight loss from initial baseline weight
DPP Class Attendance | 6 months
  Number and proportion of the classes attended
DPP Class Attendance | 12 months
  Number and proportion of the classes attended

SECONDARY OUTCOMES:
Physical Activity | 6 months
  Self-reported hours/minutes of physical activity in past week
Physical Activity | 12 months
  Self-reported hours/minutes of physical activity in past week
Blood pressure | 6 months
  Systolic and diastolic blood pressure will be measured
Blood pressure | 12 months
  Systolic and diastolic blood pressure will be measured
Blood glucose | 6 months
  Hemoglobin A1C
Blood glucose | 12 months
  Hemoglobin A1C
Office/clinic visits | 12 months
  Proportion of participants with a physician office/clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Jannette Y Berkley-Patton, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - University Health, Kansas City, Missouri
  - University of Missouri-Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided